CLINICAL TRIAL: NCT06049056
Title: Which Automated Methodology?
Acronym: WhAM
Status: Completed | Type: Observational
Sponsor: Keele University (Other)
Responsible Party: Sponsor
Other Study IDs: RG-0369-23
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Recruitment
Keywords: Primary care; Digital data collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- General Practice 1: General Practice 1 use the following methods to invite participation to the study:
  Recruitment Method 1 (RM1): Automated check-in screens containing research questions Recruitment Method 2 (RM2): SMS invites with URL link to an online questionnaire Recruitment Method 3 (RM3): Mailing containing a URL link to an online questionnaire
  Interventions: Other: Invitation
- General Practice 2: General Practice 2 use the following methods to invite participation to the study:
  Recruitment Method 1 (RM1): Automated check-in screens containing research questions Recruitment Method 2 (RM2): SMS invites with URL link to an online questionnaire Recruitment Method 3 (RM3): Mailing containing a URL link to an online questionnaire
  Interventions: Other: Invitation
- General Practice 3: General Practice 3 use the following methods to invite participation to the study:
  Recruitment Method 1 (RM1): Automated check-in screens containing research questions Recruitment Method 2 (RM2): SMS invites with URL link to an online questionnaire Recruitment Method 3 (RM3): Mailing containing a URL link to an online questionnaire
  Interventions: Other: Invitation
- General Practice 4: General Practice 4 use the following methods to invite participation to the study:
  Recruitment Method 1 (RM1): Automated check-in screens containing research questions Recruitment Method 2 (RM2): SMS invites with URL link to an online questionnaire Recruitment Method 3 (RM3): Mailing containing a URL link to an online questionnaire
  Interventions: Other: Invitation
- General Practice 5: General Practice 5 use the following methods to invite participation to the study:
  Recruitment Method 1 (RM1): Automated check-in screens containing research questions Recruitment Method 2 (RM2): SMS invites with URL link to an online questionnaire Recruitment Method 3 (RM3): Mailing containing a QR code providing access to an online questionnaire
  Interventions: Other: Invitation
- General Practice 6: General Practice 6 use the following methods to invite participation to the study:
  Recruitment Method 1 (RM1): Automated check-in screens containing research questions Recruitment Method 2 (RM2): SMS invites with URL link to an online questionnaire Recruitment Method 3 (RM3): Mailing containing a QR code providing access to an online questionnaire
  Interventions: Other: Invitation
- General Practice 7: General Practice 7 use the following methods to invite participation to the study:
  Recruitment Method 1 (RM1): Automated check-in screens containing research questions Recruitment Method 2 (RM2): SMS invites with URL link to an online questionnaire Recruitment Method 3 (RM3): Mailing containing a QR code providing access to an online questionnaire
  Interventions: Other: Invitation
- General Practice 8: General Practice 8 use the following methods to invite participation to the study:
  Recruitment Method 1 (RM1): Automated check-in screens containing research questions Recruitment Method 2 (RM2): SMS invites with URL link to an online questionnaire Recruitment Method 3 (RM3): Mailing containing a QR code providing access to an online questionnaire
  Interventions: Other: Invitation
- General Practice 9: General Practice 9 use the following methods to invite participation to the study:
  Recruitment Method 1 (RM1): Automated check-in screens containing research questions Recruitment Method 2 (RM2): SMS invites with URL link to an online questionnaire Recruitment Method 3 (RM3): Mailing containing a URL link and a QR code providing access to an online questionnaire
  Interventions: Other: Invitation
- General Practice 10: General Practice 10 use the following methods to invite participation to the study:
  Recruitment Method 1 (RM1): Automated check-in screens containing research questions Recruitment Method 2 (RM2): SMS invites with URL link to an online questionnaire Recruitment Method 3 (RM3): Mailing containing a URL link and a QR code providing access to an online questionnaire
  Interventions: Other: Invitation

INTERVENTIONS:
Other: Invitation — During Recruitment Method 3, x4 practices will send letters with a URL link providing the potential participant with access to the online questionnaire, x4 practices will send letters with a QR code providing the potential participant with access to the online questionnaire, and x2 practices will send letters with a URL link and a QR code providing the potential participant with access to the online questionnaire,

SUMMARY:
The aim of this study is to identify the modes of clinical research invitation that optimise digital responses from participants in primary care settings. This will be achieved by investigating and characterising response rates (recruitment) obtained from a hybrid of digital recruitment methods, in general practice settings.

Responses to this research will provide a single data item on general health to further characterise the sample and whether, since Covid-19, adults are more or less willing to participate in research.

DETAILED DESCRIPTION:
When conducting research, which data collection method to use, can be a difficult decision for many researchers. Choosing an inappropriate method can result in untrustworthy findings and therefore wrong conclusions. The use of digital technologies to improve the quality and reduce the cost of health care services, is a vision set out by government in 2021. How digital technologies can be used, in carrying out health research, is an area that there is not a lot known about and needs further research. This study will therefore investigate how to invite people to take part in research and which digital methods people use, to take part.

It is commonly known that the recruitment of research participants from primary care settings is difficult. The Covid-19 pandemic however highlighted the importance of primary care, in the delivery of healthcare research, which is the setting where most patients visit. Being contacted about a research study of importance, is the first step in a patients journey towards taking part in a research study. Patients will though, often drop out before they actually consent to take part in a research study. A recent NIHR survey suggested a positive increase in the public's attitude to health research. This research study will also investigate whether, since Covid-19, people are actually more or less willing to take part in research and their reasons for this.

The digital methods used for collecting data in this study, will include: automated check-in screens; Short Messaging Service (SMS or text message) with online data collection; and postal invitations from the general practice, with online data collection accessed by a quick response (QR) code or website. All people of age 18 years and over, registered at a participating general practice, will be allowed to take part. Data collected will include demographics, a data item on general health and one on willingness to take part in research.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or over.
* Adults registered at participating general practices.

Exclusion Criteria:

* People under the age of 18 years.
* Adults who have asked for their medical records not to be used for research and have a relevant code indicating this included on their records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults of age 18 years and over, registered at a participating general practice, will be eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 8880 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Recruitment (RM1) | 14 days
  Number of participants recruited to the WhAM study following receipt of an invitation to participate from an automated check-in-screen.
Recruitment (RM2) | 14 Days
  Number of participants recruited to the WhAM study following receipt of an invitation to participate from an SMS sent from the general practice.
Recruitment (RM3a) | 14 days
  Number of participants recruited to the WhAM study following receipt of an invitation to participate from an invitation letter sent from the general practice containing a QR code.
Recruitment (RM3b) | 14 days
  Number of participants recruited to the WhAM study following receipt of an invitation to participate from an invitation letter sent from the general practice containing a URL link.

SECONDARY OUTCOMES:
Willingness to participate in research since the COVID-19 pandemic | 14 days
  Number of adults that are less willing to participate in research since the Covid-19 pandemic.
Willingness to participate in research since the COVID-19 pandemic | 14 days
  Number of adults that are more willing to participate in research since the Covid-19 pandemic.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Lawton, Principal Investigator — Keele CTU
Locations (1):
- NIHR CRN: West Midlands, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No identifiable data will be collected